CLINICAL TRIAL: NCT03755076
Title: Perceptual-motor Interaction to Improve Bimanual Coordination After Stroke
Acronym: Bimanual
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: University of Pennsylvania (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Shailesh Kantak, Institute Scientist, Albert Einstein Healthcare Network
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1 R01 HD095992-01A1; R01HD092481 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-11-27 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will perform bilateral arm movements in a virtual reality environment under different perceptual conditions to identify a condition that improves coordination between arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurotypical Control (Experimental): Neurotypical healthy age-matched controls.
  Interventions: Behavioral: Perceptual cuing
- Stroke survivor (Experimental): Stroke survivors with mild-to-moderate motor impairments
  Interventions: Behavioral: Perceptual cuing

INTERVENTIONS:
Behavioral: Perceptual cuing — Participants were provided four perceptual cues (or feedback) in a pseudorandom order: (a) indiscriminate, (b) Altered gain, (c) Coordination, (d) Dual: altered gain and coordination

SUMMARY:
Significant difficulty in incorporating the weaker arm in daily activities after stroke is, in part, driven by difficulty in engaging both arms interactively in a coordinated manner.

The current study aims to determine the nature of bimanual coordination deficits after stroke and takes initial steps to test a novel theory-driven approach to improve interactive bimanual coordination in patients with stroke. This project will advance stroke rehabilitation by identifying novel, scientifically-based strategies to improve the engagement of the weaker arm in coordinated and interactive bimanual actions of daily life, thus improving quality of life in individuals after stroke.

DETAILED DESCRIPTION:
Specific Aim: Determine the immediate effects of perceptual cues on bimanual coordination in stroke survivors.

Rationale: Bimanual performance after stroke is impaired and demonstrate two principal deficits: (a) impaired spatiotemporal coordination between the two arms and (b) reduced engagement of the paretic arm. Perceptual cuing often overrides motor execution constraints to influence bimanual coordination in healthy individuals, and help improve performance. Our aim is to determine the immediate effects of specific perceptual cues on bimanual coordination in common-goal bimanual action in participants with stroke. The perceptual cue conditions are (a) indiscriminate: no specific feedback, (b) altered gain: paretic arm gain was reduced such that the paretic arm had to contribute more compared to the nonparetic arm, (c) coordination cue provided as feedback of the horizontal tilt of the common goal, (d) Dual: altered gain of the paretic arm combined with the coordination cue. Our working hypothesis is that time-lag feedback will constrain the two arms to move simultaneously, shorten the time-lag and increase CCr. Further, greater movement weighting applied to the weaker arm to increase the engagement of the weaker arm toward the bimanual action may impair bimanual coordination immediately.

Overall materials and methods: The proposed experiments will follow the general pattern we have used in previous behavioral psychophysical studies in individuals with and without stroke. A controlled virtual environment that records kinematics of the arm and allows real-time movement interaction with a virtual motor task will be used. A program integrating motion capture system (Acsention Technology TrakSTAR) and MATLAB-based GUI-gaming environment allows tracking of the two arms, experimenter-control for specific manipulation such as position of the virtual brick, target gap, relative contribution of the arms and mapping of each arm movement to the movement of the virtual brick to provide real-time and post-response feedback. Participants will be seated in an adjustable chair facing a computer monitor with their trunk constrained to the chair. Their arms will be completely supported on a low friction table top and free to move in the horizontal (X-Y) plane with minimal resistance. An opaque screen will occlude participants' direct vision of their arms. Magnetic markers will be secured to their hands just proximal to the wrist joint and the position of the markers mapped to a virtual brick shown on the computer screen. The motor task is to move the virtual brick(s) to a virtual target gap(s) on the computer screen by moving both arms in 2D (X-Y) plane on the low-friction table. While real-time visual feedback of the brick is available, the brick cannot be felt haptically. From a perceptual perspective, in independent goal condition, each arm moves its own virtual brick to the target gap. In common-goal condition, a common brick was moved on the computer screen to a target window by predetermined weighting of each arm movement.

Prior to beginning the experiments, participants will reach with the paretic arm in three different directions (135º, 90º and 45º relative to the horizontal) to record the maximum reaching distance for two trials in each direction. The minimum reach distance across the three directions will be used to calibrate the start and end position of the target gaps. The target window position will be placed at 90% of the maximum reach distance, oriented at 90º relative to the horizontal.

Procedures: Participants will come to the laboratory for a baseline evaluation to determine eligibility to participate in the experimental protocol. During this baseline evaluation, we will perform the following tests: (1) Fugl-Meyer Examination, (2) Mini-mental scale, (3) Tests for hemineglect using a line-bisection test, (4) Western Aphasia Battery for patients with Aphasia (5) TMS safety questionnaire, (6) MRI safety questionnaire, (7) Box and Block test as well as (8) Penn Neurocognitive assessment.

In the present study, we will test the effect of two different perceptual cues on bimanual coordination. Participants will be instructed to "move" a common virtual brick with both arms to the target windows at 90 degree position without tilting the brick within a target MT of 800 milliseconds- 1.2 seconds. Participants will complete four 60-trial blocks a pseudorandom order. Each block will consist 60 trials of a distinct perceptual cueing condition depending upon the nature of perceptual cues provided.

Condition 1: Indiscriminate: This condition will be similar to the common-goal bimanual condition in Aim 1 where they will transport a common virtual block fixed in a horizontal position to three targets in pseudorandom order. The movement of the bar will be an unweighted average of the two arm movements; i.e., each arm will contribute to 50% of the virtual bar movement (50-50 weighting).

Condition 2: Altered gain: This condition will be similar to Condition 1 (block fixed in horizontal position), but the arm weighting will be differential. The paretic arm will have reduced gain such that it will have to move farther to move the virtual brick with this cue than without it.

Condition 3: Coordination cue: the weighting coefficients of the two arms will be equal (i.e. 50-50); and the virtual brick will tilt in the direction of the lagging arm proportional to the relative time-lag between arms. Operational definition of relative time-lag: Relative time-lag is different than absolute time lag. Relative time-lagis the time-lag between the relative timing of each arm within its trajectory. To illustrate, if the left and right arm are contributing to 70 and 30% of the brick movement, relative time-lag at mid-movement will be zero if the left and right arm have covered half of their respective trajectories. Therefore, relative time-lag is influenced by temporal as well as spatial component of the movement of each arm. Concurrent and post-response feedback about the tilt and path of the virtual brick will be provided after each trial.

Condition 4: Dual cues combining altered gain with coordination cue: In addition to the coordination cue (i.e. "tilt" feedback about the relative time-lag), the paretic arm will have reduced gain such that it will have to move farther and faster to keep the virtual brick horizontal.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of unilateral stroke
2. ability to reach along a diagonal direction at least 80% of their arm length while fully supported on a frictionless surface and trunk constrained.
3. Mini-mental scale score > 26, OR s score of 4 or above on auditory verbal comprehension part of the Western Aphasia Battery to ensure intact comprehension and following commands.

(e) no evidence of hemispatial neglect tested by a line bisection test.

Exclusion Criteria:

1. bilateral stroke,
2. complete paralyses,
3. basal ganglia/cerebellar stroke,
4. pain or stiffness in upper extremity that will interfere with the task or inability to follow task instructions.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shailesh S Kantak, PhD, PT, Principal Investigator — Moss Rehabilitation Research Institute
Locations (1):
- Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with stroke (n=50) and age matched controls (n=29) were recruited from Moss Rehabilitation Research Registry in Pennsylvannia, PA. Recruitment occurred between April 2019- January 2024.
Pre-assignment Details: No participants were excluded from the study after enrollment.
Groups:
- Stroke Survivors: Stroke survivors with mild-to-moderate motor impairments
Period: Overall Study
Arm/Group | Neurotypical Control | Stroke Survivors
Started | 29 | 50
Condition 1:Indiscriminate | 29 | 50
Condition 2: Altered Gain | 29 | 50
Condition 3: Coordination Cue | 29 | 50
Condition 4: Dual Cues | 29 | 50
Completed | 29 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurotypical Control | Stroke Survivors | Total
Number analyzed (Participants) | 29 | 50 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.82 (10.91) | 60.52 (8.94) | 61.73 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 15 | 30 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 50 | 79
Upper Extremity Fugl-Meyer Score; Motor impairment [Mean (Standard Deviation); unit: units on a scale] — Fugl-Meyer Assessment (FMA) scale is an index to assess motor impairment of the upper extremity after stroke. The total scale ranges from 0-66; reported values are total scores. Higher scores indicate less impairment and lower scores indicate greater motor impairment.
  units on a scale | 66 (0) | 51.5 (13.45) | 56.82 (12.77)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Cross-correlation Coefficient
Description: Cross-correlation between tangential velocity profiles of the two hands was used to index spatial and temporal coordination between hands. Cross-correlation measures similarities of two distinct time series as a function of the displacement of one relative to the other. Repeated correlations between the two hand velocity profiles were obtained as the velocity profile of one hand was successively lagged. The maximum cross correlation coefficient obtained gave a measure of similarity between the two profiles, indexing spatial coordination. The better the arms moved in space, the higher the score they got, called the cross-correlation coefficient (CCr). CCr values range from zero to 1; with values close to 1 means the arms were moving very well together.
Time Frame: After 20 minutes of training under each perceptual cue condition
Measure: Mean (Standard Deviation); unit: cross-correlation coefficient
Arm/Group | Neurotypical Control | Stroke Survivors
Number analyzed (Participants) | 29 | 50
cross-correlation coefficient
  Condition 1: Indiscriminate-Baseline | 0.989 (0.014) | 0.945 (0.064)
  Condition 1: Indiscriminate-End of practice | 0.995 (.006) | 0.996 (.005)
  Condition 2: Altered gain- Baseline | 0.985 (0.016) | 0.951 (0.05)
  Condition 2: Altered gain: End of practice | 0.998 (0.003) | 0.997 (0.003)
  Condition 3: Coordination: Baseline | 0.957 (0.068) | 0.933 (0.065)
  Condition 3: Coordination: End of practice | 0.998 (0.002) | 0.995 (0.006)
  Condition 4: Dual: Baseline | 0.873 (0.184) | 0.861 (0.097)
  Condition 4: Dual: End of practice | 0.997 (0.003) | 0.990 (0.018)
Statistical Analysis 1: Comparison: Neurotypical Control vs Stroke Survivors; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Between Hands Time-lag
Description: Temporal coordination is about how well both arms move at the same time. Temporal coordination was quantified as the time lag at which the peak cross-correlation coefficient was obtained via cross-correlation analysis. If one arm moves a little later than the other, there's a time delay (or time lag). Shorter the delay, the better the timing between the arms. If the delay is positive, it means the weaker or less-used arm is moving after the stronger one.
Time Frame: After 20 minutes of training under each perceptual cue condition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Neurotypical Control | Stroke Survivors
Number analyzed (Participants) | 29 | 50
milliseconds
  Condition 1: Indiscriminate: Baseline | 19.57 (24.04) | 72.75 (149.08)
  Condition 1: Indiscriminate: End of Practice | 0.35 (0.95) | 1.55 (7.59)
  Condition 2: Altered gain: Baseline | 15.92 (18.31) | 51.51 (64.83)
  Condition 2: Altered gain: End of Practice | 0.42 (1.25) | 0.04 (0.29)
  Condition 3: Coordination: Baseline | 28.64 (27.06) | 49.15 (48.81)
  Condition 3: Coordination: End of Practice | 0.21 (1.13) | 8.44 (19.49)
  Condition 4: Dual: Baseline | 107.85 (121.29) | 152.44 (188.30)
  Condition 4: Dual: End of Practice | 0.071 (0.377) | 26.48 (76.15)
Statistical Analysis 1: Comparison: Neurotypical Control vs Stroke Survivors; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: Two days of practice
Description: The definition of adverse events did not differ from the one used in the clinicaltrials.gov.
Groups:
- Neurotypical Controls: Neurotypical healthy age-matched controls
- Stroke Survivors: Stroke survivors with mild-to-moderate impairments
Arm/Group | Neurotypical Controls | Stroke Survivors
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/50
Other Adverse Events (participants affected / at risk) | 0/29 | 0/50

LIMITATIONS AND CAVEATS:
The study included moving a virtual brick without any haptic feedback. The virtual object was used to ensure systematic manipulation of perceptual cues at this early phase of translational research. Thus future studies need to determine if these findings may be applicable in real-world tasks. We included individuals with mild-to-moderate impairments; thus, these findings may not apply to those with more severe motor and cognitive impairments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT03755076/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03755076/ICF_001.pdf